CLINICAL TRIAL: NCT01638819
Title: A Randomized, Blinded, Placebo-controlled, Crossover Study to Assess the Efficacy of Stem Cells From Autologous Umbilical Cord Blood to Improve Language and Behavior in Children With Autism
Brief Title: Autologous Cord Blood Stem Cells for Autism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sutter Health (Other)
Responsible Party: Principal Investigator, Michael Chez, MD, Principal Investigator, Sutter Health
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CB2011Chez
Record Dates: First submitted 2012-06-26; First posted 2012-07-12 (Estimated); Results first posted 2018-08-20 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Autism
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Autologous Cord Blood Stem Cells (Experimental)
  Interventions: Biological: Autologous Cord Blood Stem Cells
- Placebo (Placebo Comparator): Saline
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Autologous Cord Blood Stem Cells — One infusion of 60 ml syringe of study product
  Arms: Autologous Cord Blood Stem Cells
Biological: Placebo — Saline
  Arms: Placebo

SUMMARY:
Evaluate the efficacy of one infusion of stem cells from autologous umbilical cord blood in patients with autism over six months after infusion as measured by changes in expressive and receptive language.

Also demonstrate improved behavior, learning, and changes in Serum tumor necrosis factor alpha (TNF-α), tumor necrosis factor beta (TNF-β), interleukin 1-alpha (IL-1α), interleukin 1-beta (IL-1β), interleukin 6 (IL-6), interleukin 10 (IL-10), and interleukin 13 (IL-13).

DETAILED DESCRIPTION:
This is a single-center, randomized, placebo-controlled, crossover outpatient study with 15 subjects receiving one infusion of autologous umbilical cord blood (AUCB) containing a minimum of 10 million total nucleated cells per kilogram (TNC/kg) and 15 subjects receiving an infusion of placebo (saline). After the 24-week follow-up testing is conducted, the groups will crossover so that patients who initially received AUCB will receive placebo and patients who received placebo at baseline will receive the cord blood. Both groups will be tested again 24-weeks after infusion. The neuropsychologist, PI, staff from Cord Blood Registry (CBR), and parents will be blinded as to the infusion sequence.

The duration of participation for each study subject is approximately 55 weeks. This includes one screening visit over a period of approximately 6 weeks, one visit for baseline testing, one day for infusion of TNC (minimum 10 million/kg) or saline placebo followed by 24 weeks of follow-up. A second baseline visit is conducted at week-24 with the second infusion of TNC or saline placebo occurring 5-7 days after. Twenty-four additional weeks of follow-up occur after the second infusion.

ELIGIBILITY:
Inclusion Criteria:

* Age 2 to 7 years of age
* Diagnosis of Autistic Disorder as diagnosed by the Diagnostic and Statistical Manual, 4th Edition, Text Revision (DSM-IV-TR) developmental delays, and ADOS
* A sufficient quantity of autologous cord blood stored at Cord Blood Registry that was stored and processed using the Thermogenesis AutoXpress Platform
* Stable on any current medications for at least 2 months prior to infusion of cord blood
* Medical records indicating that patient does not have genetic conditions such as cerebral palsy, cystic fibrosis, muscular dystrophy, crohns disease, rheumatoid disease, fragile X, Retts Syndrome, Angelman Syndrome, tuberous sclerosis, epilepsy, or known genetic defects that overlap autism spectrum.
* Results of an EEG within 12-months of baseline
* English speaking

Exclusion Criteria:

* CNS infection
* Extreme prematurity (< 34 weeks gestation)
* Severe Cognitive Disability IQ below 45 with autism
* Clinical seizure activity within 6 months of baseline
* Lennox Gastaut syndrome or infantile spasms
* Dravet syndrome
* HIV, renal or hepatic impairment
* Prior hematological or malignant disease
* Fever of 101 F within 2 weeks prior to infusion
* Serious CNS infection or trauma
* Unwilling to commit to follow-up
* Mental illness including schizophrenia
* Pervasive Developmental Disorder-Not Otherwise Specified
* Asperger's Disorder
* Cord blood unit is less than 85% viable, has a TNC of less than 10 million/kg, or sterility testing results are positive
* Garlic allergy
* Previous adverse reaction to Dimethyl Sulfoxide (DMSO)
* Maternal medical records indicate communicable diseases including HIV, Hepatitis B or C, syphilis, cytomegalovirus (CMV)
* Currently taking anti-inflammatory medications
* History of asthma who may potentially require treatment with steroids
* Inflammatory Disease
* Renal/hepatic disease: serum Creatinine > 1.5 mg/dl and total Bilirubin > 1.5 mg/dl
* Allergic to diphenhydramine (Benadryl)
* Treatment with chelation therapy, hyperbaric oxygen therapy, pig worm therapy, or other alternative therapies the investigator deems clinically relevant

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2012-08; Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Chez, MD, Principal Investigator — Sutter Health
Locations (1):
- Sutter Pediatric Neurology, Sacramento, California, United States

REFERENCES:
- [Derived] Mauron A. [Autism, stem cells, and magical powder]. Rev Med Suisse. 2012 Sep 19;8(354):1795. No abstract available. French. PMID 23097920
- See also: Sutter Institute for Medical Research — http://www.checksutterfirst.org/research/

RESULTS

PARTICIPANT FLOW:
Groups:
- Autologous Cord Blood Stem Cells First/Placebo Second; Placebo First/Autologous Cord Blood Stem Cells Second: Autologous Cord Blood Stem Cells: One infusion of 60 ml syringe of study product
  Placebo: Saline
Period: Overall Study
Arm/Group | Autologous Cord Blood Stem Cells First/Placebo Second | Placebo First/Autologous Cord Blood Stem Cells Second
Started | 15 | 15
First Intervention (8 Weeks) | 15 | 15
Second Intervention (24 Weeks) | 14 | 15
Completed | 14 | 15
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Autologous Cord Blood Stem Cells First/Placebo Second | Placebo First/Autologous Cord Blood Stem Cells Second | Total
Number analyzed (Participants) | 14 | 15 | 29
Age, Continuous [Mean (Full Range); unit: years] | 4.50 [2.42 to 6.80] | 4.57 [3.00 to 6.30] | 4.53 [2.42 to 6.80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 11 | 14 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 11 | 13 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 12 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 14 | 15 | 29
Abnormal EEG at baseline [Count of Participants; unit: Participants] | 5 | 4 | 9
Autism Diagnostic Observation Schedule (ADOS) [Mean (Standard Deviation); unit: units on a scale] — The Autism Diagnostic Observation Schedule (ADOS) is a semi-structured assessment of communication, social interaction, and play (or imaginative use of materials) for individuals suspected of having autism or other pervasive developmental disorders. The total score ranges from 0 to 28 with 0 representing no abnormality present. A child is suspected to have Autism if the total ADOS score is greater than 7. The mean of the total ADOS scores is listed below.
  units on a scale | 7.93 (1.39) | 6.60 (3.14) | 7.24 (2.50)
Compartment infused [Count of Participants; unit: Participants] — Each subject's cord blood unit consists of two compartments. One contains 80% total volume and the other contains 20% total volume.
  Participants
    Large compartment (80%) | 9 | 12 | 21
    Small compartment (20%) | 5 | 3 | 8
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 19.79 (4.44) | 18.67 (3.02) | 19.21 (3.75)
TNC dose infused x 10^6/kg [Mean (Standard Deviation); unit: Number of cells infused x 10^6/kg] — The Total Nucleated Cell count or TNC is the total cell count after cord blood processing. Population: TNC data was not available for 2 cord blood first subjects and 5 placebo first subjects.
  Number of cells infused x 10^6/kg
    number analyzed (Participants) | 12 | 10 | 22
    (all) | 14.49 (6.12) | 18.17 (8.30) | 16.16 (7.26)
Viable total nucleated cell (vTNC) count infused [Mean (Standard Deviation); unit: number of alive cells x 10^6/kg] — The viable Total Nucleated Cell count or vTNC is the count of alive cells. Population: TNC dose data was not available for 2 cord blood first subjects and 5 placebo first subjects.
  number of alive cells x 10^6/kg
    number analyzed (Participants) | 12 | 10 | 22
    (all) | 314.88 (236.52) | 359.34 (163.22) | 335.09 (203.06)
Percent viability post-thaw, (flow cytometry 7-AAD) [Mean (Standard Deviation); unit: Percent viable cells] — This measure determines the percent of stem cells that are alive.
  Percent viable cells | 51.36 (11.36) | 55.75 (11.38) | 53.73 (11.37)
Percent viable CD34 (cluster of differentiation) - post-thaw [Mean (Standard Deviation); unit: Percent viable cells] — CD34, a protein found on the surface of stem cells, is the best known marker for blood-forming stem cells. It is used to predict the quality of white cell count yield.
  Percent viable cells | 49.54 (36.66) | 45.06 (37.46) | 47.30 (36.41)

OUTCOME MEASURES:

1. Primary Outcome: Change in Language (Total Standard Score, Range 40 - 160)
Description: Change in language as measured by the Receptive One-Word Vocabulary Test (ROWVT-4) and Expressive One-Word Vocabulary Test (EOWVT-4) at baseline and six months following infusion of stem cells from AUCB or infusion of placebo.
  The ROWPVT-4 and EOWPVT-4 were administered by a neuropsychologist and are norm-referenced assessments. The ROWPVT-4 tests an individual's ability to match a spoken word with an image of an object, action, or concept. The EOWPVT-4 tests an individual's ability to name, with one word, objects, actions, and concepts when presented with color illustrations. The tests target the ability to understand the meaning of words spoken and name what is depicted on a test plate without context.
  Scores of 85-115 are considered to be within the average range of functioning.
Time Frame: Baseline and 6 months
Population: Please note that endpoints for only the first 24 weeks were recorded due to the fact that the placebo second group may not be a true placebo group (stem cell infusion does not necessarily wash out like a drug).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Autologous Cord Blood Stem Cells | Placebo
Number analyzed (Participants) | 14 | 15
units on a scale
  ROWPVT-4 baseline | 79.62 (25.85) | 79.66 (21.21)
  ROWPVT-4 6 months | 80.45 (22.07) | 80.59 (26.33)
  EOWPVT-4 baseline | 74.55 (23.23) | 73.10 (20.88)
  EOWPVT-4 6 months | 74.03 (22.00) | 75.38 (23.22)

2. Secondary Outcome: Change in Behavior/Learning (Standard Score, Range 40 - 160 for Each Subtest)
Description: Change in the Vineland Adaptive Behavior and Socialization Scales (2nd edition) between baseline and six months after infusion of AUCB containing stem cells.
  Vineland Adaptive Behavior and Socialization Scales consist of the following subparts: Daily Living Skills, Socialization, and Adaptive Behavior Composite (ABC). These are questionnaires completed by a parent or caregiver. Scores above 80 are classified using approximately the same ranges as IQ tests. Scores below 80 are categorized as borderline adaptive functioning (70-80); mildly deficient adaptive functioning (51-69); moderately deficient adaptive behavior (36-50); severely deficient adaptive behavior; (20-35); and markedly or profoundly deficient adaptive behavior (<20).
Time Frame: Baseline and 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Autologous Cord Blood Stem Cells | Placebo
Number analyzed (Participants) | 14 | 15
units on a scale
  ABC - baseline | 66.00 (12.20) | 74.27 (16.00)
  ABC - 6 month | 67.57 (16.52) | 75.00 (11.60)
  Communication - baseline | 66.00 (15.56) | 79.60 (17.18)
  Communication - 6 month | 68.00 (18.82) | 83.33 (15.46)
  Motor - baseline | 73.86 (13.17) | 77.67 (13.57)
  Motor - 6 month | 69.71 (15.10) | 76.67 (7.61)
  Daily - baseline | 68.14 (15.55) | 77.13 (16.61)
  Daily - 6 month | 70.36 (17.73) | 77.33 (15.30)

3. Secondary Outcome: Change in Knowledge and Fluid Reasoning (Scaled Score, Range 1-19 for Each Subtest)
Description: The Stanford Binet, version 5, was used to assess the brain function. It can assess the level of intelligence across several age spans and ability levels. The Stanford-Binet looks at intelligence in five areas. In this study 2 areas were looked at: Knowledge and Fluid Reasoning that were age and condition appropriate. Each sub-test has a mean of 10 and a standard deviation of 3. The standard deviation indicates how far above or below the norm the subject's score is. Scores of 7 to 13 are considered to be within the average range of functioning.
Time Frame: Baseline and 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Autologous Cord Blood Stem Cells | Placebo
Number analyzed (Participants) | 14 | 15
units on a scale
  Fluid Reasoning - baseline | 5.86 (5.46) | 5.97 (5.28)
  Fluid Reasoning - 6 months | 6.79 (5.75) | 6.41 (5.69)
  Knowledge - baseline | 3.97 (3.46) | 4.45 (3.63)
  Knowledge - 6 months | 4.62 (3.75) | 4.41 (3.70)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the entire study time frame (12 months).
Description: Adverse events were measured for all participants throughout the study and not classified by arm since both arms received stem cell cord blood infusion.
Groups:
- All Participants: Adverse events were measured for all participants throughout the study and not by arm since both arms received stem cell cord blood infusion.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 28/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=29)
Seasonal cold (Respiratory, thoracic and mediastinal disorders) | 12 (18)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dark urine (Renal and urinary disorders) | 9 (9)
Flu (General disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 6 (9)
Fever (General disorders) | 13 (15)
Strep infection (Infections and infestations) | 3 (4)
Upper respiratory infection (Infections and infestations) | 3 (3)
Vomiting (Gastrointestinal disorders) | 11 (17)
Loose stool (Gastrointestinal disorders) | 1 (1)
Mononucleosis (General disorders) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Scarlet fever (Infections and infestations) | 1 (1)
Sinus infection (Infections and infestations) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Ear infection (Ear and labyrinth disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes